CLINICAL TRIAL: NCT00688233
Title: Phase 1 Effect of the Innovated Seifi's Functional Appliance on the Skeletal and Dentoalveolar Changes of Class II/Division 1, Deep Bite Cases
Brief Title: Effect of the Innovated Seifi's Functional Appliance on Skeletal and Dentoalveolar Changes of Class II/ 1, Deep Bite
Acronym: Seifi-Fx
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Professor Massoud Seifi, Shahid Beheshti Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 234567
Record Dates: First submitted 2008-05-23; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Orthodontic Appliance Design; Retrognathism; Malocclusion, Angle Class II; Deepbite
Keywords: Seifi's Functional, Class II/1, Mandibular Retrognathism
MeSH Terms: conditions — Retrognathia; Malocclusion, Angle Class II

ARMS (1):
- F-seifi (Experimental)
  Interventions: Device: Seifi's Functional

INTERVENTIONS:
Device: Seifi's Functional — Patient with Class II Division 1 and Deepbite malocclusion will wear the Seifi's Functional to get the benefit of skeletal and dentoalveolar correction.
  Other Names: Functional Therapy; Class II correction; Deepbite correction

SUMMARY:
For improving the appearance of protruded upper front teeth when lower front teeth may touch palatal mucosa or have proximity to that; the innovated Seifi's Functional Appliance may be used.

DETAILED DESCRIPTION:
Records will be obtained for each patient by the same operator before treatment and at the end of treatment. The appliance in this study is designed by Prof. Seifi and will be constructed by a well trained technician in the orthodontic laboratory of shahid Beheshti School of dentistry under the supervision of the operator. The appliance consists of a jack screw in the midpalatal region plus two Adams' clasps on the upper 1st molars and four Kimia clasps on the buccal embrasure of the upper deciduous molars or premolars. For the mandibular portion there is an incisal clasp and incisors are capped by acrylic.

The participants will be advised to use the appliance 24 hours per day except for meal times and when brushing the teeth or reading Farsi or English in class room.

Each patient will pay his/her first recall visit to the orthodontic department one week after the appliance delivery and will be instructed to turn the maxillary expansion jack screw 1:4 turn twice a week to achieve coordination of the upper and lower arches in the transverse dimension. The patients will be evaluated over one month intervals and necessary adjustments were made.

All cephalometric records, before and after treatment, will be coded and analyzed by a second party and the ultimate results and evaluations will be made.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 - 12 years old
* Class Π division 1 malocclusion (ANB>4)
* Increased over jet (>4mm)
* Increased overbite (>4mm)

Exclusion Criteria:

* History of previous orthodontic treatment
* Evidence of craniofacial syndromes

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-10 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Overjet and Overbite | 2-6 month depending on the amount of OJ and OB and the patient compliances

SECONDARY OUTCOMES:
sagittal and vertical cephalometric measurements | before-after

CONTACTS AND LOCATIONS:
Overall Officials: Massoud Seifi, DDS, MSD, Study Chair — Shahid Beheshti Medical Sciences University
Locations (1):
- Dental School, Shahid Beheshti Medical Sciences University, Tehran, Tehran Province, Iran